CLINICAL TRIAL: NCT07337317
Title: Frequency of Contrast Enhancement on Stairways
Brief Title: Evaluating Stairway Designs for Individuals With Vision Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Alabama in Huntsville (Other)
Responsible Party: Principal Investigator, Sara Harper, Assistant Professor, The University of Alabama in Huntsville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0011
Record Dates: First submitted 2025-12-19; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Vision, Low; Mobility Limitation
Keywords: older adults; impaired contrast sensivity
MeSH Terms: conditions — Vision, Low; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Four contrast frequency conditions by two lighting conditions (N = 8) will be evaluated. The four frequencies are (1) contrast markings added to all steps, (2) contrast markings added to the first, last step, (3) contrast markings added to the first, two and last, two steps, (4) no contrast markings on stairs, in both low light and standard lighting conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will participate in the experimental arm, that involves a factorial model approach inwhich all participants will experience all eight conditions.
  Interventions: Other: Frequency of contrast marking on stair steps

INTERVENTIONS:
Other: Frequency of contrast marking on stair steps — Frequency of contrast marking on stair steps will be evaluated to determine how foot clearance, perceptions in older adults with and without impaired contrast sensivity

SUMMARY:
The goal of this study is to learn if contrast frequency on step tread-edges influences foot clearance measures, a marker of fall risk, in older adults with and without visual impairments.

The main questions that aim to be answered are how foot clearance measures change across different frequencies of stair contrast, and how experiences and perceptions of different stair contrast frequencies are evaluated.

Researchers will compare individuals with and without visual impairments to see if contrast frequency on step tread-edges changes.

Participants will attend one visit during which their vision will be measured, and they will be asked to ascend and descend laboratory stairs at different contrast frequencies.

An optional second visit will entail a focus group meeting to better understand how contrast affects mobility in their home and everyday life.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ Contrast sensitivity log 1.6 or greater
2. travels independently in the community, including stairways > two times/week
3. comfortable ascending and descending a stairway with rest time provided

   Exclusion Criteria:
4. severe rheumatologic and or orthopedic diseases (e.g., awaiting joint replacement, active inflammatory disease)
5. lower-limb injuries and/or recent joint replacements (e.g., hip fracture, hip, or knee replacement within six months of study enrollment)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Toe clearance | visit 1, through study completion, an average of 1 year
  Toe, foot vertical clearance on stair steps
Heel clearance | visit 1, through study completion, an average of 1 year
  heel, foot horizontal clearance on stair steps
Frequency of <5mm toe clearances | visit 1, through study completion, an average of 1 year
  how often <5mm toe clearances occur
Frequency of <5mm heel clearances | visit 1, through study completion, an average of 1 year
  how often <5mm toe clearances occur

SECONDARY OUTCOMES:
Likert-Scale responses of contrast marking frequency conditions | visit 1, through study completion, an average of 1 year
  5-point range from strongly dislike to strongly like
Perception responses of contrast marking frequency conditions | visit 1, through study completion, an average of 1 year
  Collected via auditory responses

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Harper, PhD, Principal Investigator — University of Alabama in Huntsville
Locations (1):
- University of Alabama in Huntsville, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
We will archive our deidentified metadata to the Inter-University Consortium for Political and Social Research (ICPSR).
Supporting Information: Study Protocol, Analytic Code
Time Frame: The IDP will be made available within 6 months after publication, and will be made publicly available for 3 years.
Access Criteria: Access will be monitored through ICPSR.
URL: https://www.openicpsr.org/openicpsr/